CLINICAL TRIAL: NCT01846637
Title: Comparative Study Between Two and Five cm Resection During Laparoscopic Sleeve Gastrectomy
Brief Title: Two or Five cm From Pylorus During Laparoscopic Sleeve Gastrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ahmed Abdel-Raouf El-Geidie, assistant professor of general surgery, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2013
Record Dates: First submitted 2013-02-10; First posted 2013-05-03 (Estimated); Last update posted 2013-05-06 (Estimated); Status verified 2013-05

CONDITIONS: Morbid Obesity
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- 2 cm from pylorus (Experimental): at laparoscopic sleeve gastrectomy the distal point of gastric division is 2 cm from the pylorus.
  Interventions: Procedure: laparoscopic sleeve gastrectomy
- 6 cm from pylorus (Active Comparator): at laparoscopic sleeve gastrectomy the distal point of gastric division is 6 cm from the pylorus
  Interventions: Procedure: laparoscopic sleeve gastrectomy

INTERVENTIONS:
Procedure: laparoscopic sleeve gastrectomy

SUMMARY:
The investigators compare two techniques for laparoscopic sleeve gastrectomy. in the first one the distal margin of stapling is 2 cm from the pylorus and in the second it is 6 cm away from the pylorus.

ELIGIBILITY:
Inclusion Criteria:

* morbid obese patients

Exclusion Criteria:

* contraindication to laparoscopy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-06; Primary Completion 2013-04 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
percentage of excess weight loss | 2 years

SECONDARY OUTCOMES:
complications | 2 years

OTHER OUTCOMES:
improvement of comorbidities | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Gastroenterology Surgical Center, Al Mansurah, Dakahlia Governorate, Egypt